CLINICAL TRIAL: NCT00876824
Title: A Prospective, Multicentric, Randomized, Two Arm, Open Label Phase III Study To Assess Efficacy And Safety Of Infusion Of Amphomul® (Amphotericin B Emulsion) As Compared To Liposomal Amphotericin In Patients Of Visceral Leishmaniasis (Kala Azar)
Brief Title: To Study the Effect Of Single Infusions Of Amphotericin B Lipid Preparations in Treatment of Patients Of Kala Azar
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bharat Serums and Vaccines Limited (Industry)
Collaborators: Ministry of Science and Technology (Ambiguous)
Responsible Party: Dr. Gautam V. Daftary, Bharat Serums and Vaccines Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSV-AMBE III-KA-0908
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Leishmaniasis, Visceral
Keywords: Black Fever; Kala-Azar; Amphotericin B lipid emulsion; Liposomal Amphotericin B
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amphotericin B lipid emulsion (Experimental): Amphotericin B lipid emulsion (Amphomul) 15 mg/kg on day 1 in group A Drug: Amphotericin B lipid emulsion
  Interventions: Drug: Amphotericin B Lipid emulsion
- Liposomal Amphotericin B (Active Comparator): Liposomal Amphotericin B in visceral leishmaniasis - 15mg/kg on day 1 in Group B
  Interventions: Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B Lipid emulsion — Amphotericin B lipid emulsion (Amphomul) 15 mg/kg on day 1 in group A for treatment of Visceral Leishmaniasis
  Other Names: Amphomul
  Arms: Amphotericin B lipid emulsion
Drug: Liposomal Amphotericin B — Liposomal Amphotericin B in visceral leishmaniasis - 15 mg/kg on day 1 in group B
  Other Names: AmBisome
  Arms: Liposomal Amphotericin B

SUMMARY:
The purpose of this study is to determine whether a single bolus of dose of Amphoterin B lipid emulsion (Amphomul) is as efficacious and safe compared to a single dose Liposomal Amphotericin B in treating patients with Indian Visceral Leishmaniasis (Kala Azar).

DETAILED DESCRIPTION:
Visceral Leishmaniasis, which is progressive and fatal if not treated, is an insidious, chronic disease that is characterized by irregular fever, anorexia, weight loss, cough, gross enlargement of the spleen and liver, mild anemia and emaciation. This may be preceded by rigors and vomiting. If untreated, Kala-azar, which is the most severe form of Leishmaniasis, has a mortality rate of nearly 100%.

The goal of the project is to establish that a single dose of AMPHOMUL® can be used to achieve a Definitive cure for Visceral Leishmaniasis leading to a short course therapy. The project will also seek to establish that AMPHOMUL ® is safe, at least as effective and more affordable than current treatment, and is without the risk of drug resistance.

The trial is a Prospective, Multicentric, Randomized, Two Arm, Open label Phase III study to Assess Efficacy and Safety of Infusion of Amphomul® (Amphotericin B Emulsion) as Compared to Liposomal Amphotericin B in Patients of Visceral Leishmaniasis (Kala azar)who are either treatment naive or treatment resistant to other antileishmanial drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 5 to 65 years (both inclusive).
* Clinical signs and symptoms of Visceral Leishmaniasis (fever of over 2 weeks duration and splenomegaly)
* Presence of amastigotes (Leishmania-Donovani bodies) at prescreening detected by rK39 dipstick test with confirmation by splenic or bone marrow aspirate smear examination.
* Non-pregnant, non-lactating females of age ≥5 years, and woman of childbearing potential who are willing to use acceptable methods of contraception
* Negative Urine pregnancy test (UPT) in all women

Exclusion Criteria:

* Patients with past history of treatment with Amphotericin B or any other drug for Visceral Leishmaniasis within 30 days prior to screening.
* Patients positive for HIV, HCV and HBsAg infection, immunocompromised patients (through history).
* Concurrent diabetes, tuberculosis or bacterial pneumonia or any other infectious or major psychiatric disease.
* Pregnant or nursing women
* Patients receiving any of the medications prohibited by the study protocol.
* Simultaneous participation in another trial or received any IP <30 days prior to enrolment.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Clinical and parasitological cure at end of treatment and final cure (no relapse) at six months | Six months after dose administration

SECONDARY OUTCOMES:
To assess the Number of AEs, SAEs, Incidence of IRTs, with no Incidence of nephrotoxicity and hepatotoxicity and no change in the Laboratory values for different parameters | within 30 to 45 days from drug administration and continue throughout duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gautam Daftary, MBBS, Principal Investigator — Bharat Serums and Vaccines Ltd
Locations (2):
- India (2):
  - Muzaffarpur, Bihar
  - Patna, Bihar

REFERENCES:
- [Derived] Sundar S, Pandey K, Thakur CP, Jha TK, Das VN, Verma N, Lal CS, Verma D, Alam S, Das P. Efficacy and safety of amphotericin B emulsion versus liposomal formulation in Indian patients with visceral leishmaniasis: a randomized, open-label study. PLoS Negl Trop Dis. 2014 Sep 18;8(9):e3169. doi: 10.1371/journal.pntd.0003169. eCollection 2014 Sep. PMID 25233346